CLINICAL TRIAL: NCT01696682
Title: Study on the Difference of Anastomotic Leakage Ratio Between Wide and Narrow Gastric Conduit During Minimally Invasive Esophagectomy
Brief Title: The Optimal Width of Gastric Conduit for Minimally Invasive Esophagectomy: Wide or Narrow?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Tan, Lijie, Associate Professor of Surgery; Vice Chief, Division of Thoracic Surgery, Fudan University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ZSchest2012001
Record Dates: First submitted 2012-09-22; First posted 2012-10-01 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Anastomotic Leakage
Keywords: minimally invasive esophagectomy; anastomotic leakage; gastric conduit
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrow Gastric Conduit (Experimental): The group in which narrowed gastric conduit will be performed during minimally invasive esophagectomy
  Interventions: Procedure: Narrowed Gastric Conduit
- Wide Gastric Conduit (Experimental): The group in which widened gastric conduit will be performed during minimally invasive esophagectomy
  Interventions: Procedure: Widened Gastric Conduit

INTERVENTIONS:
Procedure: Narrowed Gastric Conduit — The gastric conduit will be formed much narrower in the intervention arm during minimally invasive esophagectomy
  Other Names: Narrowed Gastric Tube
  Arms: Narrow Gastric Conduit
Procedure: Widened Gastric Conduit — A widened gastric tube will be formed during the surgery
  Other Names: Wide Gastric Tube
  Arms: Wide Gastric Conduit

SUMMARY:
The study hypothesized that a narrow gastric conduit(less than 3cm in width) would minimize anastomotic leakage following minimally invasive esophagectomy. Therefore we raise this random-controlled research, and investigate the leakage ratio from different widths of gastric conduit formed during the operation.

DETAILED DESCRIPTION:
Patients underwent minimally invasive esophagectomy in Zhongshan Hospital of Fudan University will be enrolled and be assigned to wide or narrow gastric conduit group randomly. Intra-operative blood supply and vascular SaO2 will be observed during the operation, and the rate of anastomotic leakage, together with its clinical details will be recorded in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent minimally invasive esophagectomy(three-hole procedure)
2. Clinical Staged T1-3N0M0 esophageal cancer patients or: patients who were restaged as T1-3N0M0 esophageal cancer after neo-adjuvant therapy

Exclusion Criteria:

1. With previous cancer history
2. Severe Co-morbidity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The anastomotic leakage rate | the anastomotic leakage of participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The anastomotic leakage is a severe complication following minimally invasive esophagectomy. The definition of anastomotic leakage is determined as per the STS (SOCIETY OF THORACIC SURGEONS) database.

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, MD, Study Director — Fudan University
Locations (1):
- Division of Thoracic Surgery, Zhongshan Hospital of Fudan University, Shanghai, China